CLINICAL TRIAL: NCT06002490
Title: A Phase III b, Single-arm, Multicenter, Optimal Dose Finding Study to Assess the Efficacy and Safety of P1101 in Japanese Patients With Polycythemia Vera (PV).
Brief Title: A Study to Evaluate P1101 in Japanese PV Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaEssentia Japan K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A23-301
Record Dates: First submitted 2023-07-31; First posted 2023-08-21 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Polycythemia Vera (PV)
Keywords: Myeloproliferative Neoplasms
MeSH Terms: conditions — Polycythemia Vera; Myeloproliferative Disorders | interventions — Aspirin; Phlebotomy

STUDY DESIGN:
Intervention Model Description: Conventional treatment based on phlebotomies, low-dose aspirin (acetylsalicylic acid, 75-150 mg/day) plus the subcutaneous administration of P1101 (ropeginterferon alfa-2b) once every 2 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- P1101 (Experimental): Conventional treatment based on phlebotomies, low-dose aspirin (acetylsalicylic acid, 75-150 mg/day) plus the subcutaneous administration of pegylated proline-interferon alpha-2b (P1101, ropeginterferon alfa-2b) once every 2 weeks.
  Interventions: Drug: P1101; Drug: Low-dose aspirin; Procedure: Phlebotomy

INTERVENTIONS:
Drug: P1101 — The subjects will be treated with P1101(ropeginterferon alfa-2b), starting at a dose of 250 micrograms. The dose of P1101 will be increased to 350 micrograms 2 weeks later and to 500 micrograms another 2 weeks later, and then P1101 will be administered at a fixed dose of 500 micrograms throughout the treatment period. Although the dose may be reduced to the prior dose for reasons related to the safety or tolerability, the increased dose should be preferably maintained throughout the treatment period.
  The dose of P1101 will be increased or decreased appropriately depending on the pathological condition in the range up to 500 micrograms.
  Other Names: Ropeginterferon alfa-2b
Drug: Low-dose aspirin — Low-dose aspirin (acetylsalicylic acid) (75-150 mg/day) will be given as background therapy during the 12 months of study treatment, unless contraindicated.
  Other Names: Low-doaw Acetylsalicylic acid
Procedure: Phlebotomy — Phlebotomy is performed aiming at a hematocrit < 45%. When the hematocrit value is 45% or higher, phlebotomy is performed. The volume of phlebotomy per procedure should be 200 to 400 mL while monitoring the circulatory dynamics such as blood pressure and pulse. In the elderly and patients with cardiovascular disorders, a small volume (100-200 mL) should be considered to avoid rapid changes in hemodynamics.

SUMMARY:
This is a Phase 3 single arm study to investigate efficacy and safety of P1101's rapid titration for adult Japanese patients with PV.

DETAILED DESCRIPTION:
Eligible patients will be treated with P1101, starting at 250 μg. A starting dose of P1101 is 250 mcg, an intermediate dose is 350 mcg, and a target dose is 500 mcg. As such, subjects will not be exposed to below optimal doses within the first 4 weeks. The maximum recommended single dose is 500 μg injected every two weeks.

A primary efficacy endpoint is the rate of phlebotomy-free complete hematologic response (CHR) at Week 24, where CHR is defined as the proportion of patients who have achieved a CHR and have not required phlebotomy in the previous 12 weeks. A responder for the primary endpoint is defined as meeting all of the following criteria at Week 24: Hct (<45%), WBC (≤10 x 10^9/L), and PLT (≤400 x 10^9/L).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years old at the time of informed consent to participate in the study
2. Patients diagnosed with PV according to the WHO 2008 or 2016 criteria
3. Patients with PV who have the inadequate response to an existing therapy or whom the existing therapy is inappropriate to apply (see Appendix 6)
4. Patients with adequate hepatic function at screening defined as total bilirubin ≤1.5 x upper limit of normal (ULN), international normalized ratio (INR) of prothrombin time (PT) ≤1.5 x ULN, albumin >3.5 g/dL, alanine aminotransferase (ALT) ≤2.0 x ULN, and aspartate aminotransferase (AST) ≤2.0 x ULN.
5. Patients with hemoglobin (HGB) ≥10 g/dL in female and ≥11 g/dL in male at screening
6. Patients with a neutrophil count ≥1.5 x 10^9/L at screening
7. Patients with serum creatinine ≤1.5 x ULN at screening
8. Males, and females of childbearing potential, as well as all women <2 years after the onset of menopause, must agree to use an acceptable form of birth control until 14 days following the last dose of the study drug. Also, women must agree not to breastfeed during the study (see Appendix 4 for details)
9. Written informed consent has been obtained from the patient or the patient's legally authorized representative, and the patient is capable of complying with the study requirements.

Exclusion Criteria:

1. Patients with contraindications to or hypersensitivity to IFN-α
2. Patients with previous use of IFN-α, or previous treatment with ruxolitinib
3. Patients with comorbidity with severe or serious condition that, in the opinion of the Investigator, may impact the patient's participation in the study
4. Patients with a history of major organ transplantation
5. Pregnant or lactating females
6. Patients with any other medical condition that, in the opinion of the Investigator, might impair the outcome of the study or compliance with the requirements of the protocol. These diseases include, but are not limited to, the following:

   6.1 Patients with a history or presence of autoimmune thyroid dysfunction (clinical symptoms of hyper- or hypo-thyroidism), except late stages cases on the oral thyroid substitution therapy, where potential exacerbation under interferon therapy will not constitute any further harm to the patient 6.2 Patients with any documented history of autoimmune disease (for example, hepatitis, idiopathic thrombocytopenic purpura [ITP], scleroderma, psoriasis, or autoimmune arthritis) 6.3 Patients with clinically relevant pulmonary infiltrates, infectious pneumonia or noninfectious pneumonia at screening, or a history of interstitial pulmonary disease.

   6.4 Patients with active infection with systemic symptoms (for example, bacterial, fungal, hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infection at screening).

   6.5 Patients with any evidence of severe retinal disease (e.g., cytomegalovirus [CMV] retinitis, macular degeneration) or clinically relevant ophthalmologic disease (due to diabetes mellitus or hypertension) based on the ophthalmological assessment by specialists.

   6.6 Patients with uncontrolled depression in the opinion of the Investigator 6.7 Patients with a history of suicide attempts or at risk for suicide at screening 6.8 Patients with uncontrolled diabetes mellitus (baseline HbA1c >7%) 6.9 Patients with active thromboembolism or active abdominal bleeding due to PV 6.10 Patients with a history of malignancy within the last 5 years [excluding adequately treated non-melanoma skin cancers, post-prostatectomy prostate-specific antigen (PSA) failure, healed cervical intraepithelial neoplasia and ductal carcinoma in situ (DCIS), stage 1 endometrial carcinoma, or solid tumors (without myelopathy), including other lymphomas that have not had evidence of disease for at least 2 years after treatment].

   6.11 Patients with a history of alcohol or drug abuse within the recent one year 6.12 Patients with a history or evidence of post-polycythemia vera myelofibrosis (post-PV MF), essential thrombocythemia, or MPN other than PV
7. Patients who received any other study treatment or concomitant medication with other study drug within 4 weeks prior to the first dose of study drug in this study or not recovered from any prior exposure to any other study drug.
8. Patients with symptomatic splenomegaly
9. Patients with circulating blasts in the peripheral blood within the last 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Proportion of Subjects Who Achieved Durable Phlebotomy-free Complete Hematological Response (CHR) at Week 24 | 24 weeks

SECONDARY OUTCOMES:
Rate of achieving "phlebotomy-free complete hematologic response (CHR)" (the same criteria as for the primary efficacy endpoint) at both Week 12 and Week 24. | Week12, Week24
Time to achieve CHR | Up to Week24
Time to reach response maintenance dose (three consecutive doses of the same dose) | Up to Week24
Numbers of phlebotomy required and changes in numbers of phlebotomy required from baseline | Baseline, up to Week24
Time to first response in peripheral blood count (Hct, WBC, and PLT) | Up to Week24
Duration of response in peripheral blood count (Hct, WBC, and PLT) | Up to Week24
Improvement of symptoms assessed by MPN-SAF TSS at each visit | Up to Week24
  Rated on a scale of 0-10 on an 11-point scale, with 0 being no symptoms, 1 being the best, and 10 being the worst.
Proportion of subjects without thrombotic or hemorrhagic events at Weeks 12 and 24 | Week12, week24
Change from baseline to Week 24 in JAK2 V617F allele burden level | Baseline, week24
Collect and measure Pharmacokinetics (PK) at trough | Day1, Week2, Week4, Week6, Week8, Week10, Week12, Week14, Week16, Week18, Week20, Week22, Week24

CONTACTS AND LOCATIONS:
Locations (6):
- Japan (6):
  - Mie University Hospital, Mie
  - Osaka University Hospital, Osaka
  - Kansai Medical University Hospital, Osaka
  - Juntendo University Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - University of Yamanashi Hospital, Yamanashi